CLINICAL TRIAL: NCT01236729
Title: The Effects of Primary Knee Replacement for Osteoarthritis on Disability in Activities of Daily Living and Self-rated Health in Older People
Brief Title: Disability and Self-rated Health Following Primary Knee Replacement
Status: Completed | Type: Observational
Sponsor: Coxa, Hospital for Joint Replacement (Other)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Esa Jamsen, MD, PhD, Researcher, Coxa, Hospital for Joint Replacement
Other Study IDs: KL122009
Record Dates: First submitted 2009-12-22; First posted 2010-11-09 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis; Knee Replacement
Keywords: knee replacement; disability; older people
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee replacement recipients: Patients (aged 75 years or over) with late-stage arthritis who have undergone or are undergoing primary knee replacement

SUMMARY:
Knee replacement is an effective treatment in late-stage osteoarthritis. It reduces pain and improves quality of life. There is, however, limited data concerning its results in older people and on its effect on how patients survive in regular activities of daily living (ADL), such as bathing and shopping. In this study, the results of knee replacement are evaluated from the point of view of disability in everyday activities and self-rated health. Moreover, association with ADL performance and clinical knee scores and severity of osteoarthritis are assessed.

DETAILED DESCRIPTION:
This is a cross-sectional study with a 12 month follow-up for recruited patients. Most data are gathered by a postal questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age 75 years or more at the time of operation
* diagnosis of knee osteoarthritis
* scheduled for or operated on with primary knee replacement

Exclusion Criteria:

* died during the follow-up
* inflammatory arthritides

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients refererred to or operated on with primary knee replacement in a population-based tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2009-12; Primary Completion 2013-11-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Disability in activities of daily living | Baseline (recruitment) and at 12 months

SECONDARY OUTCOMES:
Overall self-rated health | Baseline (recruitment) and at 12 months
Health-related quality of life (WOMAC) | Baseline and 12 months postoperatively
  For patients recruited in 2011-2012.

CONTACTS AND LOCATIONS:
Overall Officials: Esa Jämsen, MD, PhD, Study Director — Coxa, Hospital for Joint Replacement
Locations (1):
- Coxa, Hospital for Joint Replacement, Tampere, Finland

REFERENCES:
- [Result] Limnell K, Jamsen E, Huhtala H, Jantti P, Puolakka T, Jylha M. Functional ability, mobility, and pain before and after knee replacement in patients aged 75 and older: a cross-sectional study. Aging Clin Exp Res. 2012 Dec;24(6):699-706. doi: 10.3275/8718. Epub 2012 Nov 12. PMID 23147559
- [Result] Vekama L, Puolakka T, Honkasalo M, Huhtala H, Moilanen T, Jamsen E. Functional gain following knee replacement in patients aged 75 and older: a prospective follow-up study. Aging Clin Exp Res. 2015 Dec;27(6):865-76. doi: 10.1007/s40520-015-0348-x. Epub 2015 Mar 24. PMID 25800623